CLINICAL TRIAL: NCT02408965
Title: A Randomized Controlled Trial of Methylergonovine Prophylaxis After Dilation and Evacuation Abortion
Brief Title: Uterotonic Prophylaxis Trial
Acronym: UPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UP Trial 2015
Record Dates: First submitted 2015-03-11; First posted 2015-04-06 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — Methylergonovine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methergine (Experimental): Methergine group 0.2 mg of methylergonovine maleate single injection when manual cervical dilation begins the day before the procedure
  Interventions: Drug: Methergine
- saline placebo (Placebo Comparator): Placebo group saline single injection when manual cervical dilation begins the day before the procedure
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Methergine — 0.2 mg of methylergonovine maleate
  Other Names: methylergonovine maleate
  Arms: methergine
Other: placebo — saline placebo to maintain blinding
  Arms: saline placebo

SUMMARY:
Excessive bleeding after dilation and evacuation (D&E) requiring interventions is common, occurring in approximately 30% of cases at one large abortion-providing clinic. Uterotonic prophylaxis at the time of D&E, particularly with methylergonovine maleate (MM), is a common practice among D&E providers despite nearly no evidence for its efficacy. Finding ways to decrease excessive bleeding after D&E has the potential both to improve patient safety and to reduce costs of provider-initiated interventions. The investigators propose a randomized, controlled trial to investigate the efficacy of MM prophylaxis versus placebo in decreasing excessive bleeding measured by a composite outcome among women undergoing D&E at 20 to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 wks 0 days gestation and 24 wks 0 days gestation
* English or Spanish speaking
* BP before injection 140/90 or below
* 18 years old or over

Exclusion criteria:

* hypertension either on the preoperative or operative day (defined as systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg)
* D&E procedures with more than one day of cervical preparation with dilators
* use of protease inhibitors
* known coagulopathy
* known morbidly adherent placenta

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kerns, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- SFGH Women's Options Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Determined ineligible (n=28) Patient withdrew (n=6) Administrative error (n=2)
Groups:
- Methergine: Methergine group
- Placebo: Placebo group
Period: Overall Study
Arm/Group | Methergine | Placebo
Started | 140 | 144
Completed | 140 | 144
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methergine | Placebo | Total
Number analyzed (Participants) | 140 | 144 | 284
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24.5 [21 to 29] | 25 [21 to 31] | 24.8 [21 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 144 | 284
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic white | 39 | 48 | 87
  Non-Hispanic black | 26 | 33 | 59
  Hispanic | 37 | 33 | 70
  Asian | 7 | 7 | 14
  Mixed | 19 | 15 | 34
  Other | 11 | 8 | 19
Body mass index [Median (Inter-Quartile Range); unit: kg/m2] | 26.5 [23 to 31] | 26 [23 to 29] | 26.3 [23 to 30]
Nulliparous [Count of Participants; unit: Participants] | 35 | 37 | 72
Prior cesarean section [Count of Participants; unit: Participants] | 24 | 27 | 51
Gestation [Median (Inter-Quartile Range); unit: weeks] | 21.6 [21 to 23] | 21.5 [20 to 23] | 21.6 [20 to 23]
Needed mechanical dilation [Count of Participants; unit: Participants] | 7 | 5 | 12
Length of procedure [Median (Inter-Quartile Range); unit: minutes] | 12 [8 to 16] | 12 [9 to 15] | 12 [8 to 15]
Procedural measured blood loss [Median (Inter-Quartile Range); unit: mL] | 300 [150 to 400] | 250 [150 to 425] | 275 [150 to 410]
Current or recent cocaine or methamphetamine use [Count of Participants; unit: Participants] | 11 | 19 | 30
History of bleeding disorder [Count of Participants; unit: Participants] | 2 | 3 | 5
Preoperative systolic BP [Mean (Standard Deviation); unit: mmHg] | 112 (11) | 112 (10) | 112 (10)
Preoperative diastolic BP [Mean (Standard Deviation); unit: mmHg] | 68 (9) | 69 (8) | 69 (8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Excessive Bleeding as Determined by the Composite Outcome Criteria
Description: Clinical factors included in composite outcome of excessive bleeding after D&E:
  Post-procedure total blood loss > 125cc (after D&E) Transfusion Admission for bleeding Re-aspiration for bleeding Balloon tamponade Uterine artery embolization Major surgery for bleeding At least 1 uterotonic medication given Prescription given for any uterotonic medication at discharge Uterine compression (uterine massage or manual pressure for 2 minutes
Time Frame: Approximately 1-2 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Methergine | Placebo
Number analyzed (Participants) | 140 | 144
Participants | 78 | 75
Statistical Analysis 1: Comparison: Methergine vs Placebo; Test type: Superiority; p = 0.5, Chi-squared

2. Primary Outcome: Amount of Post-procedure Blood Loss Measured in mL
Description: post-procedure blood loss measured in recovery room
Time Frame: measured 1 to 2 hours after procedure
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Methergine | Placebo
Number analyzed (Participants) | 140 | 144
mL | 126 [86 to 166] | 76 [65 to 88]
Statistical Analysis 1: Comparison: Methergine vs Placebo; Test type: Superiority; p = 0.02, t-test, 2 sided

3. Primary Outcome: Number of Participants Who Had a Balloon Tamponade Placed From Start of Procedure to Hospital Discharge
Description: number of participants who had a balloon tamponade placed
Time Frame: duration of procedure and until discharged from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Methergine | Placebo
Number analyzed (Participants) | 140 | 144
Participants | 20 | 10
Statistical Analysis 1: Comparison: Methergine vs Placebo; Test type: Superiority; p = 0.04, Chi-squared

4. Primary Outcome: Number of Participants Who Returned to OR for Re-aspiration During Recovery Period
Description: Returned to OR for re-aspiration
Time Frame: from cervical preparation through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Methergine | Placebo
Number analyzed (Participants) | 140 | 144
Participants | 4 | 0
Statistical Analysis 1: Comparison: Methergine vs Placebo; Test type: Superiority; p = 0.06, Chi-squared

5. Primary Outcome: Number of Participants Who Were Admitted for Bleeding After Procedure
Description: hospital admission for bleeding post-procedure
Time Frame: post-procedure and during recovery until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Methergine | Placebo
Number analyzed (Participants) | 140 | 144
Participants | 4 | 0
Statistical Analysis 1: Comparison: Methergine vs Placebo; Test type: Superiority; p = 0.06, Chi-squared

6. Primary Outcome: Number of Participants Given Any Uterotonic
Description: any uterotonic medication given intraoperative or postoperative
Time Frame: intra-operative or post-operative until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Methergine | Placebo
Number analyzed (Participants) | 140 | 144
Participants | 56 | 43
Statistical Analysis 1: Comparison: Methergine vs Placebo; Test type: Superiority; p = 0.07, Chi-squared

7. Secondary Outcome: Number of Participants Who Reported Nausea up to One Hour After Procedure
Description: Patients' completed survey regarding side effects in recovery room.
Time Frame: Assessed approximately 1 hour after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Methergine | Placebo
Number analyzed (Participants) | 140 | 144
Participants | 42 | 18
Statistical Analysis 1: Comparison: Methergine vs Placebo; Test type: Superiority; p < 0.001, Chi-squared

8. Secondary Outcome: Number of Patients Who Reported Vomiting up to One Hour After Procedure
Description: Patients' completed survey regarding side effects in recovery room.
Time Frame: Assessed approximately 1 hour after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Methergine | Placebo
Number analyzed (Participants) | 140 | 144
Participants | 18 | 8
Statistical Analysis 1: Comparison: Methergine vs Placebo; Test type: Superiority; p = 0.03, Chi-squared

9. Secondary Outcome: Number of Participants Who Reported Cramping up to One Hour After Procedure
Description: Patients' completed survey regarding side effects in recovery room.
Time Frame: Assessed approximately 1 hour after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Methergine | Placebo
Number analyzed (Participants) | 140 | 144
Participants | 100 | 84
Statistical Analysis 1: Comparison: Methergine vs Placebo; Test type: Superiority; p = 0.02, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 years, March 2015 to March 2017
Description: It took from March 2015 to March 2017 to meet the study sample size. Therefore, the timeframe March 2015 through March 2017 is the duration that adverse events were monitored/collected.
Arm/Group | Methergine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/144
Serious Adverse Events (participants affected / at risk) | 4/140 | 0/144
Other Adverse Events (participants affected / at risk) | 20/140 | 11/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methergine (N=140) | Placebo (N=144)
admission to hospital for bleeding (Reproductive system and breast disorders) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methergine (N=140) | Placebo (N=144)
Balloon tamponade (Reproductive system and breast disorders) | 20 (20) | 10 (10)
reasperation (Reproductive system and breast disorders) | 4 (4) | 1 (1)
transfusion (Reproductive system and breast disorders) | 3 (3) | 0 (0)
uterine artery embolization (Reproductive system and breast disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Designed our study using a one-sided hypothesis given our belief that methergine could not cause increased bleeding based on postpartum data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-04-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02408965/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02408965/SAP_001.pdf